CLINICAL TRIAL: NCT01353898
Title: A Multiple Dose Clinical Trial to Study the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK-1972 in HIV-1 Infected Patients
Brief Title: Study of MK-1972 in Human Immunodeficiency Virus (HIV)-1 Infected Participants Who Have Not Previously Received Antiretroviral Therapy (MK-1972-003)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1972-003; 2011-000071-14 (EudraCT Number)
Record Dates: First submitted 2011-05-12; First posted 2011-05-16 (Estimated); Results first posted 2016-02-05 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-07

CONDITIONS: HIV-1 Infection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- MK-1972 50 mg once daily (Part I) (Experimental): Ten capsules containing a total daily dose of 50 mg MK-1972 or placebo were taken orally, once per day for 10 days (Part I)
  Interventions: Drug: MK-1972; Drug: Placebo to MK-1972
- MK-1972 200 mg once daily (Part I) (Experimental): Ten capsules containing a total daily dose of 200 mg MK-1972 or placebo were taken orally, once per day for 10 days (Part I)
  Interventions: Drug: MK-1972; Drug: Placebo to MK-1972
- MK-1972 800 mg once daily (Part I) (Experimental): Ten capsules containing a total daily dose of 800 mg MK-1972 or placebo were taken orally, once per day for 10 days (Part I)
  Interventions: Drug: MK-1972; Drug: Placebo to MK-1972
- MK-1972 25 mg twice daily (Part I) (Experimental): Ten capsules containing a total daily dose of 25 mg MK-1972 or placebo were taken orally, twice per day for 10 days (Part I)
  Interventions: Drug: MK-1972; Drug: Placebo to MK-1972
- MK-1972 100 mg twice daily (Part I) (Experimental): Ten capsules containing a total daily dose of 100 mg MK-1972 or placebo were taken orally, twice per day for 10 days (Part I)
  Interventions: Drug: MK-1972; Drug: Placebo to MK-1972
- Placebo twice daily (Part I) (Placebo Comparator): Ten capsules containing placebo were taken orally, twice per day for 10 days (Part I)
  Interventions: Drug: Placebo to MK-1972
- MK-1972 800 mg twice daily (Part II) (Experimental): Ten capsules containing a total daily dose of 800 mg MK-1972 or placebo were taken orally, twice per day for 10 days (Part II)
  Interventions: Drug: MK-1972; Drug: Placebo to MK-1972
- Placebo twice daily (Part II) (Placebo Comparator): Ten capsules containing placebo were taken orally, twice per day for 10 days (Part II)
  Interventions: Drug: Placebo to MK-1972

INTERVENTIONS:
Drug: MK-1972 — MK-1972 will be supplied as 25 and 100 mg capsules, and will be given orally, at a dose dependent on the treatment arm; participants will take ten capsules (active drug and/or placebo) once or twice per day for 10 days
  Arms: MK-1972 100 mg twice daily (Part I); MK-1972 200 mg once daily (Part I); MK-1972 25 mg twice daily (Part I); MK-1972 50 mg once daily (Part I); MK-1972 800 mg once daily (Part I); MK-1972 800 mg twice daily (Part II)
Drug: Placebo to MK-1972 — Placebo will be supplied as matching 25 and 100 mg capsules, and will be given orally, at a dose dependent on the treatment arm; participants will take ten capsules (active drug and/or placebo) once or twice per day for 10 days

SUMMARY:
This is a two part study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of MK-1972 in participants with HIV-1 infections. In Part 1, participants will be randomized to receive MK-1972 (at one of 5 different dose levels given once or twice per day) or placebo. Part II will begin after the results of Part I are known; participants will be randomized to receive MK-1972 (only one dose level, twice per day) or placebo. The primary hypotheses are that MK-1972 at the studied doses is safe and well tolerated in HIV-1 infected males; and that MK-1972 has superior antiretroviral activity compared to placebo.

ELIGIBILITY:
Inclusion Criteria

* Stable baseline health.
* Appropriate use of contraception; condom protection with pregnant partners.
* Documented HIV-1 positive
* Anti-retroviral therapy (ART)-naïve, defined as having never received any antiretroviral agent or ≤30 consecutive days of an investigational antiretroviral agent, excluding an integrase inhibitor, or ≤60 consecutive days of combination ART excluding an integrase inhibitor.
* No investigational agent or licensed ART within 30 days of study drug administration.
* Diagnosis of HIV-1-infection ≥ 3 months prior to screening.

Exclusion Criteria

* History of stroke, chronic seizures, or major neurological disorder.
* History of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological (outside of HIV-1 infection), renal, respiratory, or genitourinary abnormalities or diseases.
* History of clinically significant neoplastic disease.
* Use of any immune therapy agents or immunosuppressive therapy within 1 month prior to treatment in this study.
* Requirement for chronic daily prescription medications.
* Current (active) diagnosis of acute hepatitis due to any cause.
* History of chronic Hepatitis C unless there has been documented cure and/or participant with a positive serologic test for Hepatitis C virus (HCV) has a negative HCV viral load.
* Positive Hepatitis B surface antigen.
* Refusal to stop using any medication, including prescription and non-prescription drugs or herbal remedies (such as St. John's Wort [Hypericum perforatum]) beginning approximately 2 weeks (or 5 half-lives) prior to administration of the initial dose of study drug, throughout the study (including washout intervals), until the post-study visit.
* Consumption of excessive amounts of alcohol, defined as greater than 3 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [284 mL/10 ounces], wine [125 mL/4 ounces], or distilled spirits [25 mL/1 ounce]) per day.
* Consumption of excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, or other caffeinated beverages per day.
* Smoker of more than 10 cigarettes/day unwilling to restrict smoking to ≤10 cigarettes per day.
* Major surgery, donation or loss of 1 unit of blood (approximately 500 mL) or participation in another investigational study within 4 weeks prior to screening.
* History of significant multiple and/or severe allergies (including latex allergy), or an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food.
* Current regular user of any illicit drugs or has a history of drug (including alcohol) abuse within approximately 1 year. Participants with a positive cannabis test with no evidence of drug-dependency may be enrolled at the discretion of the investigator.
* History of hepatic or gallbladder disease or history of clinically significant abnormalities in liver function tests, or history of Gilbert's Syndrome, or history of elevated unconjugated bilirubin.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-06-21 (Actual); Primary Completion 2012-01-03 (Actual); Study Completion 2012-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=1972-003&kw=1972-003&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two treatment groups planned for Part II (800 mg MK-1972 twice daily, and Placebo twice daily) were not enrolled, and are therefore not included in these Results.
Period: Overall Study
Arm/Group | MK-1972 50 mg Once Daily (Part I) | MK-1972 200 mg Once Daily (Part I) | MK-1972 800 mg Once Daily (Part I) | MK-1972 25 mg Twice Daily (Part I) | MK-1972 100 mg Twice Daily (Part I) | Placebo Twice Daily (Part I)
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Study site terminated | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-1972 50 mg Once Daily (Part I) | MK-1972 200 mg Once Daily (Part I) | MK-1972 800 mg Once Daily (Part I) | MK-1972 25 mg Twice Daily (Part I) | MK-1972 100 mg Twice Daily (Part I) | Placebo Twice Daily (Part I) | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.5 (14.8) | 24.0 (2.8) | 32.5 (0.7) | 47.5 (10.6) | 37.0 (1.4) | 37.0 (17.0) | 34.9 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 2 | 2 | 2 | 2 | 2 | 2 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Clinical and Laboratory Adverse Events (AEs)
Description: An adverse event is any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR's product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the SPONSOR's product, is also an adverse event.
Time Frame: From consent to 14 days after the last dose (up to Day 24)
Population: All participants who received at least one dose of the investigational drug, according to the treatment they actually received.
Measure: Number; unit: Participants
Arm/Group | MK-1972 50 mg Once Daily (Part I) | MK-1972 200 mg Once Daily (Part I) | MK-1972 800 mg Once Daily (Part I) | MK-1972 25 mg Twice Daily (Part I) | MK-1972 100 mg Twice Daily (Part I) | Placebo Twice Daily (Part I)
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2
Participants | 2 | 1 | 2 | 2 | 1 | 2

2. Secondary Outcome: The Area Under the Curve From 0-24 Hours (AUC0-24hrs) on Day 10 for Plasma Concentration of MK-1972 in Participants With HIV-1 Infection
Description: Plasma concentration of MK-1972 was determined from blood collected from HIV-1 infected participants on Day 10 : pre-dose up to 24 hours post-dose in order to determine the AUC0-24hrs.
Time Frame: Day 10: pre-dose, and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours post-dose
Population: All participants who comply with the protocol sufficiently to ensure that these data will be likely to exhibit the effects of treatment, according to the underlying scientific model. MK-1972 was not measured for the placebo group since it did not receive any of this drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM.hr
Arm/Group | MK-1972 50 mg Once Daily (Part I) | MK-1972 200 mg Once Daily (Part I) | MK-1972 800 mg Once Daily (Part I) | MK-1972 25 mg Twice Daily (Part I) | MK-1972 100 mg Twice Daily (Part I) | Placebo Twice Daily (Part I)
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 0
nM.hr | 1540 (24.3) | 3590 (43.8) | 12500 (15.5) | 676 (27.6) | 1800 (114) |
Statistical Analysis 1: Comparison: MK-1972 200 mg Once Daily (Part I); Compared to historical data for AUC0-24hrs measured on Day 7 for healthy participants treated with 200 mg MK-1972 once daily; Test type: Superiority or Other; Geometric Mean Ratio = 0.62 — Geometric mean ratio of HIV-1/Healthy. Analyzed using a linear mixed model with fixed factors: dose, health-status and the interaction between dose and health-status
Statistical Analysis 2: Comparison: MK-1972 800 mg Once Daily (Part I); Compared to historical data for AUC0-24hrs measured on Day 7 for healthy participants treated with 800 mg MK-1972 once daily; Test type: Superiority or Other; Geometric Mean Ratio = 0.84 — [estimate comment as in outcome 2, analysis 1]

3. Primary Outcome: Change From Baseline to Day 10 in Plasma Human Immunodeficiency Virus (HIV)-1 Ribonucleic Acid (RNA) Due to Treatment With MK-1972 or Placebo
Description: Blood was collected at baseline and on Day 10, and the plasma concentration for HIV-1 RNA was determined using the Abbott RealTime HIV assay.
Time Frame: Baseline and Day 10 (24 hours post-dose)
Population: All participants who comply with the protocol sufficiently to ensure that these data will be likely to exhibit the effects of treatment, according to the underlying scientific model.
Measure: Mean (Standard Error); unit: log10 copies/mL
Arm/Group | MK-1972 50 mg Once Daily (Part I) | MK-1972 200 mg Once Daily (Part I) | MK-1972 800 mg Once Daily (Part I) | MK-1972 25 mg Twice Daily (Part I) | MK-1972 100 mg Twice Daily (Part I) | Placebo Twice Daily (Part I)
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2
log10 copies/mL | -0.97 (0.20) | -0.60 (0.30) | -1.06 (0.60) | -0.60 (0.42) | -1.90 (0.33) | -0.07 (0.05)
Statistical Analysis 1: Comparison: MK-1972 50 mg Once Daily (Part I) vs Placebo Twice Daily (Part I); Test type: Superiority or Other; Mean Difference (Final Values) = -0.90
Statistical Analysis 2: Comparison: MK-1972 200 mg Once Daily (Part I) vs Placebo Twice Daily (Part I); Test type: Superiority or Other; Mean Difference (Final Values) = -0.54
Statistical Analysis 3: Comparison: MK-1972 800 mg Once Daily (Part I) vs Placebo Twice Daily (Part I); Test type: Superiority or Other; Mean Difference (Final Values) = -0.99
Statistical Analysis 4: Comparison: MK-1972 25 mg Twice Daily (Part I) vs Placebo Twice Daily (Part I); Test type: Superiority or Other; Mean Difference (Final Values) = -0.53
Statistical Analysis 5: Comparison: MK-1972 100 mg Twice Daily (Part I) vs Placebo Twice Daily (Part I); Test type: Superiority or Other; Mean Difference (Final Values) = -1.83

ADVERSE EVENTS:
Time Frame: Up to Day 24
Arm/Group | MK-1972 50 mg Once Daily (Part I) | MK-1972 200 mg Once Daily (Part I) | MK-1972 800 mg Once Daily (Part I) | MK-1972 25 mg Twice Daily (Part I) | MK-1972 100 mg Twice Daily (Part I) | Placebo Twice Daily (Part I)
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/2 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 1/2 | 2/2 | 2/2 | 1/2 | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-1972 50 mg Once Daily (Part I) (N=2) | MK-1972 200 mg Once Daily (Part I) (N=2) | MK-1972 800 mg Once Daily (Part I) (N=2) | MK-1972 25 mg Twice Daily (Part I) (N=2) | MK-1972 100 mg Twice Daily (Part I) (N=2) | Placebo Twice Daily (Part I) (N=2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 0 (0) | 2 (4) | 0 (0) | 1 (3) | 0 (0)
Muscle contractions involuntary (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.